CLINICAL TRIAL: NCT04862741
Title: A Randomized, Double-blind Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral NX-13 in Active Ulcerative Colitis
Brief Title: Safety, Tolerability, and Pharmacokinetics of Oral NX-13 in Active Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Landos Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NX-13-1b
Record Dates: First submitted 2021-03-10; First posted 2021-04-28 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — NX-13

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NX-13 250mg IR (Experimental): Oral
  Interventions: Drug: NX-13 250mg IR
- NX-13 500mg IR (Experimental): Oral
  Interventions: Drug: NX-13 500mg IR
- NX-13 500mg MR (Experimental): Oral
  Interventions: Drug: NX-13 500mg MR
- Placebo (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NX-13 250mg IR — Subjects will take study drug by ingesting one tablet per day, recommended at the same time in the morning for consistency. Subjects in a NX-13 group will receive either 250 mg or 500 mg of NX-13 in an immediate release or modified release tablet and subjects in the placebo group will receive matched placebo.
  Arms: NX-13 250mg IR
Drug: NX-13 500mg IR — Subjects will take study drug by ingesting one tablet per day, recommended at the same time in the morning for consistency. Subjects in a NX-13 group will receive either 250 mg or 500 mg of NX-13 in an immediate release or modified release tablet and subjects in the placebo group will receive matched placebo.
  Arms: NX-13 500mg IR
Drug: NX-13 500mg MR — Subjects will take study drug by ingesting one tablet per day, recommended at the same time in the morning for consistency. Subjects in a NX-13 group will receive either 250 mg or 500 mg of NX-13 in an immediate release or modified release tablet and subjects in the placebo group will receive matched placebo.
  Arms: NX-13 500mg MR
Drug: Placebo — Subjects will take study drug by ingesting one tablet per day, recommended at the same time in the morning for consistency. Subjects in a NX-13 group will receive either 250 mg or 500 mg of NX-13 in an immediate release or modified release tablet and subjects in the placebo group will receive matched placebo.
  Arms: Placebo

SUMMARY:
This is a Phase 1b, randomized, double-blind, multicenter dose-ranging study to evaluate the safety, tolerability, and PK of NX-13. Approximately 40 subjects will be randomized in a 3:3:3:1 ratio to receive 1 of 3 NX-13 treatment regimens (NX-13 250 mg IR, 500 mg IR, 500 mg MR) (12 evaluable subjects at each of the 3 dose levels) or placebo (4 subjects), once daily for 28 consecutive days.

DETAILED DESCRIPTION:
Following screening period (up to 28 days in length), a total of 40 subjects are planned to be enrolled into this study from multiple sites in the United States, Australia, New Zealand, and Moldova. Eligible subjects will be randomized in a 3:3:3:1 ratio to receive 1 of 3 NX-13 treatment regimens (NX-13 250 mg IR, 500 mg IR, 500 mg MR) or placebo via a computer-generated interactive web response system (IWRS). Each of the NX-13 treatment groups will comprise 12 subjects and 4 subjects will be randomized to receive placebo. The study will include a maximum of 25% of subjects who have had prior exposure to biologic therapy for UC.

Dosing will extend over a 28-day period at each dose level. Subjects will receive the first dose of study drug in clinic on Day 1 (Visit 2) and Day 28 (Visit 4/EOT) but will self-administer IP at home once daily for the remaining dosing days. The study duration will be approximately 63 days: Screening Period (28 days) + Treatment Period (28 days) + Safety Follow-up (7 days after last dose). There will be a follow-up visit on Day 35 (Visit 5).

ELIGIBILITY:
Key Inclusion Criteria:

* male and female subjects aged 18 to 75 years (inclusive) with a diagnosis of UC ≥ 90 days before screening;
* active UC defined as a total Mayo Score of 4 to 10 (inclusive), at baseline, with a Mayo endoscopic subscore (MES) ≥ 2 confirmed by a central reader;
* baseline fecal calprotectin ≥ 250 μg/g;
* biologic-naïve or having stopped biologic therapy ≥ 8 weeks before the start of the study;
* 5-aminosalicylates must be stable for ≥ 1 month prior to randomization.

Key Exclusion Criteria:

* Crohn's disease (CD), indeterminate colitis, or presence or history of fistula with CD;
* a history of toxic megacolon, abdominal abscess, symptomatic colonic stricture, or stoma;
* history of or at imminent risk of colectomy;
* history of or current colonic dysplasia ;
* recent history (within 2 years prior to randomization) or current adenomatous colonic polyps;
* treatment with an immunosuppressant within 3 months of randomization;
* bacterial or parasitic pathogenic enteric infection;
* live virus vaccination within 1 month prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events after multiple oral dose administration of NX-13 in subjects with active ulcerative colitis (UC) | 63 days
  Incidence of Treatment-Emergent Adverse Events after multiple oral dose administration of NX-13

SECONDARY OUTCOMES:
PK profile of NX-13 after multiple oral dose administration in subjects with active UC | 63 days
  NX-13 concentrations in plasma, colonic tissue biopsies, and feces
PK Parameters - Time to maximum concentration (tmax); | 63 days
  NX-13 concentrations, time to maximum concentration
PK Parameters- Maximum concentration (Cmax) | 63 days
  NX-13 concentrations, maximum concentration
PK Parameters- Area under the concentration-time curve from time 0 to last measurable time-point (AUC0-tlast); | 63 days
  NX-13 concentrations, area under the concentration-time curve from time 0 to last measurable
PK Parameters-Terminal half-life (t1/2) | 63 days
  NX-13 terminal half-life PK
PK Parameters- clearance (CL); | 63 days
  NX-13 clearance PK
PK Parameters- Vz, apparent volume of distribution during terminal phase. | 63 days
  NX-13 - Vz, apparent volume of distribution during terminal phase.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Lichtiger, MD, Study Director — Landos Biopharma Inc.
Locations (31):
- United States (22):
  - Avant Research Associates LLC, Huntsville, Alabama
  - Om Research LLC, Lancaster, California
  - Allameh Medical Corporation, Mission Viejo, California
  - California Medical Research Associates, Inc., Northridge, California
  - Clinical Research of California, Walnut Creek, California
  - I.H.S Health LLC, Kissimmee, Florida
  - University of Miami Crohn's and Colitis Center, Miami, Florida
  - Valencia Medical and Research Center, Miami, Florida
  - Care Access, Orlando, Florida
  - Gastroenterology Associates of Pensacola, P.A., Pensacola, Florida
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Care Access, New York, New York
  - Care Access, Lumberton, North Carolina
  - Optimed Research, LTD, Columbus, Ohio
  - Care Access, Pottsville, Pennsylvania
  - Galen Medical Group, Chattanooga, Tennessee
  - Avant Research Associates, LLC, Austin, Texas
  - Biopharma Informatics, LLC, Houston, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Victoria Gastroenterology, Victoria, Texas
  - Care Access Research, Salt Lake City, Salt Lake City, Utah
- Ukraine (9):
  - Communal Enterprise I.I.Mechnykov Dnipropetrovsk Regional Clinical Hospital of Dnipropetrovsk Regional Counsil, cont., Dnipro
  - Communal Non-commercial Enterprise Regional Clinical Hospital of Ivano-Frankivsk Regional Council, Ivano-Frankivsk
  - Medical Center 'Ok!Clinic+' of Copmany with limited liability "International institue of Clinical Research", Kyiv
  - Clinical Hospital "Feofaniya" of State Management of Affairs, Center of Gastroenterology and Endocrinology, Kyiv
  - Communal Non-commercial Enterprise of Kyiv Regional Council Kyiv Regional Hospital, Department of Therapy, Kyiv
  - Communal Non-Commercial Enterprise of M.I. Pyrohov Vinnytsia Regional Clinical Hospital of Vinnytsia Regional Council, Vinnytsia
  - Communal Non-commercial Enterprise Vinnytsia City Clinical Hospital #1, Department of Gastroenterology, Vinnytsia
  - Medical Center of Limited Liability Company Gastroenterology Center IBD TEAM, Zaporizhzhya
  - Communal Non-commercial Enterprise O.F. Herbachevskyi Regional Clinical Hospital of Zhytomyr Regional Council, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verstockt B, Vermeire S, Peyrin-Biroulet L, Mosig R, Feagan BG, Colombel JF, Siegmund B, Rieder F, Schreiber S, Yarur A, Panaccione R, Dubinsky M, Lichtiger S, Cataldi F, Danese S. The Safety, Tolerability, Pharmacokinetics, and Clinical Efficacy of the NLRX1 agonist NX-13 in Active Ulcerative Colitis: Results of a Phase 1b Study. J Crohns Colitis. 2024 May 31;18(5):762-772. doi: 10.1093/ecco-jcc/jjad192. PMID 37952114